CLINICAL TRIAL: NCT03477110
Title: SPARE-Scalp Preservation and Radiation Plus Alternating Electric Tumor Treatment Field (NovoTTF, Optune) for Patients With Glioblastoma: A Pilot Study
Brief Title: Temozolomide, Radiation Therapy, and Tumor Treating Fields Therapy in Treating Participants With Glioblastoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17P.346; JT 10706 (Other: JeffTrial Number)
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (temozolomide, radiation, NovoTTF-200A device) (Experimental): Participants receive temozolomide PO QD starting day 1 to the end of radiation therapy and undergo 30 fractions of radiation therapy over 15-20 minutes each, 5 days a week (Monday-Friday) for 6 weeks. Beginning day 1 of radiation therapy, participants undergo tumor treatment fields therapy using NovoTTF-200A device over 18 hours or more daily in the absence of disease progression or unacceptable toxicity. Beginning 28 days after the last dose of radiation therapy, participants receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Temozolomide; Radiation: Radiation Therapy; Device: NovoTTF-200A Device; Procedure: Tumor Treating Fields Therapy

INTERVENTIONS:
Drug: Temozolomide — Given PO
  Other Names: 362856; Temcad; Temodal; Methazolastone; Temodar
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; RT
Device: NovoTTF-200A Device — Undergo tumor treatment fields therapy using NovoTTF-200A device
  Other Names: Optune
Procedure: Tumor Treating Fields Therapy — Undergo tumor treatment fields therapy using NovoTTF-200A device
  Other Names: Alternating Electric Field Therapy

SUMMARY:
This pilot early phase I trial studies the side effects of temozolomide, radiation therapy, and tumor treating fields therapy using Novo tumor treatment fields (TTF)-200A device in participants with glioblastoma. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. NovoTTF-200A device is a portable device that produces alternating electrical fields that may disrupt growth of cancer cells. Giving temozolomide, radiation therapy, and tumor treating fields therapy using NovoTTF-200A device may work better in treating participants with glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and toxicity of combination chemoradiotherapy with NovoTTF-200A device (Optune) treatment in newly diagnosed glioblastoma.

SECONDARY OBJECTIVES:

I. To determine the median progression-free survival of patients with newly diagnosed glioblastoma treated with radiotherapy with concurrent and adjuvant temozolomide plus Optune.

II. To evaluate the median overall survival, 1-year overall survival, and event-free survival.

III. Collect tumor O(6)-Methylguanine-DNA-methyltransferase (MGMT) methylation status and isocitrate dehydrogenase (IDH) mutation status.

IV. To evaluate the level of circulating tumor deoxyribonucleic acid (DNA) in glioblastoma patient serum during treatment.

V. To evaluate the quality of life of patients treated with radiotherapy with concurrent and adjuvant temozolomide plus Optune.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathology confirmed newly diagnosed World Health Organization (WHO) grade IV glioma
* Karnofsky performance status (KPS) ≥ 60
* Patients must have recovered from the effects of surgery per treating physician's judgment; there must be a minimum of 21 days from the day of surgery to the day of protocol treatment; for core or needle biopsy, a minimum of 14 days must have elapsed prior to the day of protocol treatment
* Absolute neutrophil count (ANC) ≥ 1,000 cells/mm^3
* Platelets ≥ 100,000 cells/mm^3
* Hemoglobin ≥ 9.0 g/dl
* Creatinine clearance > 30 mL/min
* Bilirubin < 2.0 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) < 3 x upper limit of normal range
* Women of childbearing potential must have a negative beta-human chorionic gonadotropin (HCG) pregnancy test documented within 14 days prior to registration
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 4 months after last dose of temozolomide
* Is able to have magnetic resonance imaging (MRI) with contrast of the brain
* All subjects must be able to comprehend and sign a written informed consent document. If the subject can comprehend the informed consent but is unable to sign, a LAR may sign the written informed consent document.

Exclusion Criteria:

* Infratentorial disease (defined as glioblastoma [GBM] derived from cerebellum or brainstem)
* Implanted pacemaker, defibrillator or deep brain stimulator, or documented clinically significant arrhythmias
* A skull defect (such as, missing bone with no replacement)
* Women of childbearing potential who are pregnant or breastfeeding
* Evidence of increased intracranial pressure (midline shift > 5 mm, clinically significant papilledema)
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study, in the opinion of the investigator
* Prior radiation treatment to the brain
* Prior treatment with temozolomide
* Known hypersensitivity to conductive hydrogels like the gel used on electrocardiogram (ECG) stickers or transcutaneous electrical nerve stimulation (TENS) electrodes
* Known active collagen vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
NovoTTF-200A device discontinuation rate due to skin toxicity | Up to 30 days after finishing chemoradiation treatment
  Discontinuation events are defined as the discontinuation of NovoTTF-200A device for > 7 consecutive days due to skin toxicity of grade 3 or higher. For discontinuation rates, the method of Atkinson and Brown will be used to allow for the two-stage design. Descriptive analysis will be performed on the acute toxicity data.

SECONDARY OUTCOMES:
Progression-free survival | From enrollment up to 1 year
  Will be evaluated using the Kaplan-Meier method.
Overall survival | From enrollment up to 1 year
  Will be evaluated using the Kaplan-Meier method.
Event-free survival | From enrollment up to 1 year
  Will be evaluated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Wenyin Shi, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ali AS, Lombardo J, Niazi MZ, Miller RC, Alnahhas I, Martinez NL, Andrews DW, Judy KD, Shi W. Concurrent chemoradiation and Tumor Treating Fields (TTFields, 200 kHz) for patients with newly diagnosed glioblastoma: patterns of progression in a single institution pilot study. J Neurooncol. 2022 Nov;160(2):345-350. doi: 10.1007/s11060-022-04146-w. Epub 2022 Nov 10. PMID 36355259
- [Derived] Miller R, Song A, Ali A, Niazi M, Bar-Ad V, Martinez N, Glass J, Alnahhas I, Andrews D, Judy K, Evans J, Farrell C, Werner-Wasik M, Chervoneva I, Ly M, Palmer J, Liu H, Shi W. Scalp-Sparing Radiation With Concurrent Temozolomide and Tumor Treating Fields (SPARE) for Patients With Newly Diagnosed Glioblastoma. Front Oncol. 2022 Apr 29;12:896246. doi: 10.3389/fonc.2022.896246. eCollection 2022. PMID 35574391
- [Derived] Song A, Bar-Ad V, Martinez N, Glass J, Andrews DW, Judy K, Evans JJ, Farrell CJ, Werner-Wasik M, Chervoneva I, Ly M, Palmer JD, Liu H, Shi W. Initial experience with scalp sparing radiation with concurrent temozolomide and tumor treatment fields (SPARE) for patients with newly diagnosed glioblastoma. J Neurooncol. 2020 May;147(3):653-661. doi: 10.1007/s11060-020-03466-z. Epub 2020 Mar 23. PMID 32206976
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/